CLINICAL TRIAL: NCT01857986
Title: A Study to Evaluate Air Leak Detection Above the Endotracheal Cuff in Intubated Patients Using the AnapnoGuard 100 System
Brief Title: Evaluating Air Leak Detection in Intubated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospitech Respiration (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HST-AG-07
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Critical Care
Keywords: Endotracheal intubation; Mechanical ventilation; Critical care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Subjects in the study group will be connected to the AnapnoGuard 100 control unit operating in the normal clinical mode (automatic CO2 leak measurement above the cuff, cuff pressure control, evacuation of secretions and tracheal rinsing)
  Interventions: Device: AnapnoGuard 100 control unit
- Control group (Active Comparator): Subjects in the control group will be connected to the AnapnoGuard 100 control unit. In the control group, the cuff pressure control of the AnapnoGuard 100 control unit will be disabled (OFF). CO2 level above the cuff will be recorded. Suction and rinsing function will operate after the system detects no CO2.
  Interventions: Device: AnapnoGuard 100 control unit

INTERVENTIONS:
Device: AnapnoGuard 100 control unit

SUMMARY:
This trial is designed to assess the effectiveness of the AnapnoGaurd 100 system relative to standard of care (SOC) Control, in the course of mechanical ventilation and intubation. The main effectiveness aspect of this trial is the AnapnoGaurd 100's ability to reduce leaks between the endotracheal tube and the trachea walls as a result of the cuff pressure management. Since the primary outcome can't be measured by any method other than the investigational device, the study groups will be treated as follows:

* The Treatment group in this study will be treated with the fully functional AnapnoGaurd 100 device (per its intended use),
* The Control group will be treated with the AnapnoGuard device, where the cuff control will be disabled (off) and the cuff management will be done according to SOC.

Effectiveness will be measured by the duration and level of carbon dioxide (CO2) leakage around the endotracheal tube (ETT) cuff, from the lungs to the subglottic space and safety will be measured by adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 (men and women);
2. Subject is expected to receive mechanical ventilation for more than 12 hours;
3. Connection of the ETT to the AnapnoGuard system within 12 hours from intubation initiation;
4. Subject or subject's legally acceptable representative signed the Informed Consent Form

Exclusion Criteria:

1. Subjects with facial, oropharyngeal or neck trauma 2. BMI>40 3. Pregnant women 4. Patient ventilated in prone position 5. Difficult intubation (defined as more than 3 intubation attempts)

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, MD, Study Director — Hospitech Respiration; Gil Bolotin, MD, Principal Investigator
Locations (4):
- Israel (4):
  - Mayanei Hayeshua Medical Center, General ICU, Bnei Brak
  - Rambam Medical Center, Cardiac Surgery Department, Haifa
  - Rambam Medical Center, Neurosurgery Department, Haifa
  - Wolfson Medical Center, General ICU, Holon

RESULTS

PARTICIPANT FLOW:
Groups:
- Study: Study patients were connected to the AnapnoGuard 100 system, using all functional modalities: active cuff pressure control, using subglottic CO2 readings as an indicator for leaks and automatic, periodic rinsing and suction of subglottic secretions.
- Control: Control patients were connected to the AnapnoGuard 100 system, with automatic, periodical rinsing and suction of subglottic secretions, while the cuff pressure control was not active (turned OFF). In the control group, the system recorded the CO2 levels in the subglottic space, but cuff pressure was managed manually using a manometer 3 times daily.
Period: Overall Study
Arm/Group | Study | Control
Started | 39 | 37
Completed | 34 | 30
Not Completed | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study | Control | Total
Number analyzed (Participants) | 34 | 30 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (18.8) | 66.7 (11.2) | 65.8 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 23
  Male | 23 | 18 | 41

OUTCOME MEASURES:

1. Primary Outcome: CO2 Leakage Above the ETT Cuff, Measured Over Time.
Description: Trial outcome measure represents patients' exposure to CO2 leakage standardized per hour. Specifically, each patients' area under the curve (AUC) of CO2 leakage (mmHg) is computed over the whole trial by multiplying leakage duration (X-axis; continuous time) by CO2 level (Y-axis; mmHg), divided by the patient's number of hours in the trial. Outcome measure is thus [CO2 mmHg*hour]/hour.
  CO2 leakage is the concentration of CO2 above the cuff as measured by the AG100 system every few minutes (in clinical mode). Time points which created the curve were every two adjacent time intervals having a valid CO2 reading.
Time Frame: Subjects will be followed for the duration of endotracheal intubation, an expected average of 4 days
Measure: Mean (Standard Deviation); unit: [CO2 mmHg*hour]/hour
Arm/Group | Study | Control
Number analyzed (Participants) | 34 | 30
[CO2 mmHg*hour]/hour | 0.09 (0.04) | 0.22 (0.32)

2. Secondary Outcome: Number of the Cuff Pressure Measurements Within the Safety Accepted Range (24 and 40cmH2O)
Description: mean number of cuff pressure measurements within the safety accepted range of 24 and 40 cmH2O, normalized using the total number of valid cuff pressure measurements.
Time Frame: Subjects will be followed for the duration of endotracheal intubation, an expected average of 4 days
Measure: Mean (Standard Deviation); unit: normalized number of Cp measurements
Arm/Group | Study | Control
Number analyzed (Participants) | 34 | 30
normalized number of Cp measurements | 0.979 (0.064) | 0.397 (0.302)

3. Post Hoc Outcome: Duration of Significant CO2 Leakage
Description: Time (minutes) of CO2 leakage readings at or above 2 mmHg
Time Frame: Subjects will be followed for the duration of endotracheal intubation, an expected average of 4 days
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Study | Control
Number analyzed (Participants) | 34 | 30
minutes | 4.61 (3.53) | 34.53 (83.27)

ADVERSE EVENTS:
Description: Four patients enrolled into the Control group were not connected to the investigational system (i.e. the AnapnoGuard 100 system). For this reason, safety data was collected only for 33 patients and not for the total 37 patients who were enrolled into this group.
Arm/Group | Study | Control
Serious Adverse Events (participants affected / at risk) | 3/39 | 4/33
Other Adverse Events (participants affected / at risk) | 7/39 | 6/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Study (N=39) | Control (N=33)
Death (General disorders) | 3 | 3
Hemodynamic instability (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Study (N=39) | Control (N=33)
Atrial Fibrilation (Cardiac disorders) | 1 | 2
Infection of surgery wound (Infections and infestations) | 1 | 1
Melena (Gastrointestinal disorders) | 0 | 1
Massive bleeding after surgery (Injury, poisoning and procedural complications) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less